CLINICAL TRIAL: NCT02469181
Title: Impact of Enzyme Replacement Therapy on Cardiac Function in Patients With Fabry's Cardiomyopathy : A Prospective Multi-modality Imaging Study Using Diastolic Stress Echocardiography, LV Vortex Flow and Cardiac MRI(RECAFTURE Trial)
Brief Title: Impact of Enzyme Replacement Therapy on Cardiac Function in Patients With Fabry's Cardiomyopathy (RECAFTURE Trial)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0679
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Fabry's Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lyso GL-3
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FD(Fabry disease) group: 28 patients with newly diagnosed genetically confirmed Anderson-Fabry's disease will undergo diastolic stress echocardiography, LV vortex flow analysis, and cardiac MRI before enzyme replacement therapy(ERT) (baseline study) and after 1 year of treatment with agalsidese beta at the dose of 1mg/kg (follow-up study).

SUMMARY:
The purpose of this study is to evaluate the impact of ERT on LV diastolic function and flow in patients with Fabry's cardiomyopathy using diastolic stress echocardiography, LV vortex flow and CMR.

DETAILED DESCRIPTION:
1. Objectives -The purpose of this study is to evaluate the impact of ERT on LV diastolic function and flow in patients with Fabry's cardiomyopathy using diastolic stress echocardiography, LV vortex flow and CMR.
2. Primary / Secondary Endpoint 1) Primary endpoint

   * Changes of peak exercise E/E' by diastolic stress echocardiography (RECAP-F STRESS trial) and LV vortex flow parameters (RECAP-F FLOW trial) at 1 year follow up.

     2) Secondary endpoint
   * Changes of extracellular volume by CMR(T1 mapping) at 1 year follow up (RECAP-F trial) ② Evaluation of the degree of the resting LV diastolic function ③ Other echo-parameters; LV mass index at baseline, 1 year follow up, reduction of peak exercise E/E prime at 1 year follow up

     * Changes of quality of life using questionnaire ⑤ Change of peak VO2, exercise time, AT by diastolic stress echocardiography at 1 year follow up ⑥ Change in T1 baseline(myo, ms) & T1 baseline(blood, ms) T1 postcontrast(myo, ms) & T1 baseline(blood, ms) by CMR
3. Study Methods 1) Study Design : 28 patients with newly diagnosed genetically confirmed Anderson-Fabry's disease will undergo diastolic stress echocardiography, LV vortex flow analysis, and cardiac MRI before enzyme replacement therapy(ERT) (baseline study) and after 1 year of treatment with agalsidese beta at the dose of 1mg/kg (follow-up study).

2) Study procedures : Examinations as described below will be done before ERT and 1 year later

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16~75 years with Fabry's disease who were confirmed by enzyme assay and gene study
* All patients should have LV hypertrophy in 2D echocardiography (end diastolic septum and posterior wall thickness ≥12mm)
* Patients provided with the written, informed consent to participate in this study

Exclusion Criteria:

* Contraindication for agalsidase beta enzyme replacement treatment
* Patients who cannot perform supine bicycle stress echocardiography, contrast echocardiography or cardiac MRI
* Hemodynamically significant valvular heart disease or arrythmias
* History of acute myocardial infarction or congestive heart failure with reduced LV ejection fraction of less than 35%
* CVA in the prior 6 months
* Scheduled or planned surgery in the next 6 months
* Chronic liver cirrhosis
* Allergy to contrast agent (Definity®, Lantheus Medical Imaging, North Billerica, MA, USA)

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 16~75years with Fabry's disease who were confirmed by enzyme assay and gene study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-05-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Changes of peak exercise E(velocity of early)/E'(Early diastolic) by diastolic stress echocardiography | 1 year after the echocardiography

SECONDARY OUTCOMES:
Change of peak VO2 by diastolic stress echocardiography | 1 year after the echocardiography
Change of peak exercise time by diastolic stress echocardiography | 1 year after the echocardiography
LV(left ventricular) vortex flow analysis by contract echocardiography | 1 year after the echocardiography
Changes of extracellular volume by Cardiac MRI(CMR) | 1 year after the CMR

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea